CLINICAL TRIAL: NCT03041467
Title: Randomized Study of IN.PACT™ AV Access Paclitaxel-Coated Percutaneous Transluminal Angioplasty (PTA) Balloon vs. Standard PTA for the Treatment of Obstructive Lesions in the Native Arteriovenous Dialysis Fistulae (AVF)
Brief Title: IN.PACT™ AV Access IDE Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Endovascular (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: APV-IN.PACT AV Access
Record Dates: First submitted 2017-02-01; First posted 2017-02-02 (Estimated); Results first posted 2020-02-27 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2023-06

CONDITIONS: Arteriovenous Fistula Stenosis; Arteriovenous Fistula Occlusion; Arteriovenous Fistula; Fistula
MeSH Terms: conditions — Arteriovenous Fistula; Fistula

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- IN.PACT AV DCB (Experimental): PTA will be performed using the IN.PACT AV Access Drug Coated Balloon. IN.PACT AV Access DCB was the device name used during the clinical study. Medtronic has changed the name of the device to IN.PACT™ AV Paclitaxel-Coated Balloon Catheter (also referred as IN.PACT AV DCB). Hence, throughout posting, the study device will be referred to as the "IN.PACT AV DCB."
  Interventions: Device: IN.PACT AV DCB
- Standard Balloon Angioplasty (Active Comparator): PTA will be performed using a commercially available uncoated PTA balloon.
  Interventions: Device: Standard Balloon Angioplasty

INTERVENTIONS:
Device: IN.PACT AV DCB — IN.PACT™ AV Paclitaxel-Coated Percutaneous Transluminal Angioplasty (PTA) Balloon
  Arms: IN.PACT AV DCB
Device: Standard Balloon Angioplasty — Standard PTA Balloon
  Arms: Standard Balloon Angioplasty

SUMMARY:
To evaluate the safety and efficacy of the IN.PACT™ AV Access Drug Coated Balloon (DCB) compared to percutaneous transluminal angioplasty (PTA) for treatment of subjects presenting with de novo or non-stented restenotic obstructive lesion of native arteriovenous dialysis fistulae (AVF) in the upper extremity.

DETAILED DESCRIPTION:
This is a prospective, global, multi-center, single-blinded, 1:1 randomized clinical trial evaluating the IN.PACT™ AV Access Drug Coated Balloon (DCB) compared to percutaneous transluminal angioplasty (PTA) for treatment of subjects presenting with de novo or non-stented restenotic obstructive lesion of native arteriovenous dialysis fistulae (AVF) in the upper extremity. The trial will be conducted in up to 30 sites in the United States, Japan, and New Zealand.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is ≥21 years of age.
2. Patient has a life expectancy of ≥ 12 months
3. Patient has a native AV fistula created ≥ 60 days prior to the index procedure
4. The target AV fistula has undergone successful dialysis for at least 8 of 12 sessions during a four week period
5. Patient has a de novo and/or non-stented restenotic lesion located between the arteriovenous anastomosis and axillosubclavian junction with ≥50% stenosis. Note: If the lesion is located in the anastomosis, the treatment may be delivered up to 2 cm upstream on the arterial side. If the lesion is located in the cephalic arch, the treatment may be delivered up to 2 cm into the subclavian vein
6. Patient has a target lesion or a tandem lesion that is ≤ 100 mm in length (by visual estimate) Note: Tandem lesions may be enrolled provided they meet all of the following criteria: Separated by a gap of ≤ 30mm (3 cm), total combined lesion length, including 30 mm gap, ≤ 100 mm, and able to be treated as a single lesion
7. Patient has a target vessel diameter of 4.0 - 12.0 mm (by visual estimate).
8. Patient underwent successful crossing of the target lesion with the guide wire and pre-dilatation with a high pressure PTA balloon defined as: residual stenosis of ≤ 30% and absence of a flow limiting dissection (Grade ≥ C) or perforation
9. Patient provides written consent prior to enrollment in the study
10. Patient is willing to comply with all follow-up evaluations at specified times

Exclusion Criteria:

1. Women who are breastfeeding, pregnant, or are intending to become pregnant, or men intending to father children
2. Patient is receiving immunosuppressive therapy
3. Patient is anticipating a kidney transplant within 6 months of enrollment into the study
4. Patient has undergone prior intervention of access site within 30 days of index procedure
5. Patient with anticipated conversion to peritoneal dialysis
6. Patient has an infected AV access or systemic infection
7. Patient has planned surgical revision of access site
8. Patient with secondary non-target lesion requiring treatment within 30-days post index procedure
9. Patient with hemodynamically significant central venous stenoses that cannot be successfully treated prior to treatment of the target lesion
10. Patient with target AVF or access circuit which previously had or currently has a thrombosis
11. Patients judged to have a lesion that prevents complete inflation of an angioplasty balloon or proper placement of the delivery system
12. Patient with target lesion located central to the axillosubclavian junction
13. Patient has significant arterial inflow lesion requiring treatment more than 2 cm upstream from the anastomosis in the AV access
14. Patient has presence of pseudoaneurysm or aneurysm requiring treatment at the lesion site
15. Patient has presence of a stent located in the target AV access circuit
16. Patients with known allergies or sensitivities to paclitaxel
17. Patient with known contraindication, including allergic reaction, or sensitivity to contrast material that cannot be adequately pre-treated
18. Patient who cannot receive recommended antiplatelet and/or anticoagulant therapy
19. Patient with clinically significant Steal Syndrome requiring treatment
20. Patient is enrolled in another investigational drug, device, or biological study and has not completed the primary endpoint, or was previously enrolled in this study
21. Patient has a comorbid-condition that, in the judgment of the Investigator, may cause him/her to be non-compliant with the protocol of confound data interpretation

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330 (Actual)
Dates: Start 2017-04-25 (Actual); Primary Completion 2018-12-06 (Actual); Study Completion 2023-05-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Lookstein, MD, Principal Investigator — The Mount Sinai Hospital; Andrew Holden, MD, Principal Investigator — Auckland City Hospital; Hiroaki Haruguchi, MD, Principal Investigator — Haruguchi Vascular Access Clinic
Locations (29):
- United States (21):
  - University of Alabama at Birmingham (UAB) Hospital, Birmingham, Alabama
  - SKI Vascular Center, Tempe, Arizona
  - Capital Nephrology Medical Group, Sacramento, California
  - Florida Research Network, Gainesville, Florida
  - Coastal Vascular and Interventional, Pensacola, Florida
  - Christie Clinic Vein and Vascular Center, Champaign, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - King's Daughters Medical Center, Ashland, Kentucky
  - Mayo Clinic, Rochester, Minnesota
  - Holy Name Medical Center, Teaneck, New Jersey
  - The Mount Sinai Hospital, New York, New York
  - North Carolina Nephrology PA, Raleigh, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Dialysis Access Institute, Orangeburg, South Carolina
  - Sanford University of South Dakota Medical Center, Sioux Falls, South Dakota
  - University Surgical Associates, Chattanooga, Tennessee
  - Dallas Nephrology Associates, Plano, Texas
  - Sentara Vascular Specialists, Norfolk, Virginia
  - Richmond Vascular Center, North Chesterfield, Virginia
  - Vascular Institute of Virginia, Woodbridge, Virginia
- Japan (6):
  - Kansai Rosai Hospital, Amagasaki
  - Shonan Kamakura General Hospital, Kamakura
  - Kishiwada Tokushukai Hospital, Kishiwada
  - Saitama Medical Center Saitama Medical University, Saitama
  - Shizuoka General Hospital, Shizuoka
  - Tokyo Women's Medical University Hospital, Tokyo
- New Zealand (2):
  - Auckland City Hospital, Auckland
  - Capital and Coast District Health Board, Wellington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lookstein RA, Haruguchi H, Ouriel K, Weinberg I, Lei L, Cihlar S, Holden A; IN.PACT AV Access Investigators. Drug-Coated Balloons for Dysfunctional Dialysis Arteriovenous Fistulas. N Engl J Med. 2020 Aug 20;383(8):733-742. doi: 10.1056/NEJMoa1914617. PMID 32813949

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 330 subjects from 21 US sites and 8 OUS sites contributed to the global cohort. 204 of subjects came from U.S. sites, 112 of subjects came from Japan sites, and 14 of subjects came from New Zealand sites. There was no minimum enrollment requirement at each site; individual sites were not allowed to enroll more than 20% of the total study subjects.
Pre-assignment Details: A total of 488 patients were consented to be reviewed for enrollment. 158 patients were not enrolled in the study. 170 subjects were randomized to IN.PACT AV Drug Coated Balloon treatment and 160 subjects were randomized to the Standard PTA Treatment.
Groups:
- IN.PACT AV DCB: PTA will be performed using the IN.PACT AV Drug Coated Balloon.
  IN.PACT AV DCB: IN.PACT™ AV Paclitaxel-Coated Percutaneous Transluminal Angioplasty (PTA) Balloon
Period: Overall Study
Arm/Group | IN.PACT AV DCB | Standard Balloon Angioplasty
Started | 170 | 160
30 Days | 159 | 154
3 Months | 158 | 151
6 Months | 145 | 144
9 Months | 138 | 138
12 Months | 131 | 121
18 Months | 123 | 113
24 Months | 110 | 101
36 Months | 75 | 58
48 Months | 54 | 41
60 Months | 57 | 41
Completed | 57 | 41
Not Completed | 113 | 119
Not completed — Death | 46 | 39
Not completed — Withdrawal by Subject | 36 | 37
Not completed — Lost to Follow-up | 6 | 8
Not completed — Declined consent for study extension | 21 | 33
Not completed — Exit reason other than withdrawal, death, or lost to follow up | 4 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | IN.PACT AV DCB | Standard Balloon Angioplasty | Total
Number analyzed (Participants) | 170 | 160 | 330
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.8 (13.1) | 65.5 (13.4) | 65.6 (13.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 58 | 59 | 117
  Male | 112 | 101 | 213
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 42 | 46 | 88
  Black or African American | 54 | 48 | 102
  Asian | 63 | 57 | 120
  Native Hawaiian or Other Pacific Islander | 6 | 4 | 10
  American Indian or Alaska Native | 0 | 0 | 0
  Other | 5 | 5 | 10
Region of Enrollment [Number; unit: participants]
  New Zealand | 8 | 6 | 14
  United States | 104 | 100 | 204
  Japan | 58 | 54 | 112
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: 3 subjects in each treatment group did not provide data regarding ethnicity.
  Participants
    number analyzed (Participants) | 167 | 157 | 324
    Hispanic or Latino | 15 | 14 | 29
    Not Hispanic or Latino | 152 | 143 | 295

OUTCOME MEASURES:

1. Primary Outcome: Target Lesion Primary Patency Rate Through 6 Months
Description: Freedom from clinically-driven target lesion revascularization (CD-TLR) or access circuit thrombosis measured through 6 months post-procedure.
Time Frame: 6 Months Post-Procedure
Population: Evaluable subjects were all subjects with events or subjects without events but had at least 150 days of clinical follow-up were counted as evaluable subjects. If a subject had no event and abandoned AV Access circuit within 150 days the subject will be considered not evaluable for 6-months effectiveness endpoints.
Measure: Count of Participants; unit: Participants
Arm/Group | IN.PACT AV DCB | Standard Balloon Angioplasty
Number analyzed (Participants) | 152 | 148
Participants | 125 | 88
Statistical Analysis 1: Comparison: IN.PACT AV DCB vs Standard Balloon Angioplasty; Test type: Superiority; p < 0.001, One-sided Z-test

2. Primary Outcome: Primary Safety Endpoint - Serious Adverse Event Rate
Description: Serious Adverse Event (SAE) rate involving the AV access circuit
Time Frame: 30 days post procedure
Population: All subjects with events or subjects without events but had at least 23 days of clinical follow-up were counted as evaluable subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | IN.PACT AV DCB | Standard Balloon Angioplasty
Number analyzed (Participants) | 166 | 158
Participants | 7 | 7
Statistical Analysis 1: Comparison: IN.PACT AV DCB vs Standard Balloon Angioplasty; Test type: Non-Inferiority — Non-inferiority p-values for the primary safety endpoint was based on the Farrington-Manning non-inferiority test with a margin of 7.5%; p = 0.002, Farrington-Manning Test

3. Secondary Outcome: Access Circuit Primary Patency
Description: Defined as freedom from re-intervention in the access circuit or access circuit thrombosis through 3 months, 6 months, 9 months,12 months, 18 months, and 24 months post-procedure.
Time Frame: 3, 6, 9, 12, 18, and 24 Months
Population: There is no planned hypothesis test other than at 6 months time point.
Measure: Number; unit: Percentage of participants
Groups:
- IN.PACT AV DCB: PTA was performed using the IN.PACT AV Drug Coated Balloon.
  IN.PACT AV DCB: IN.PACT™ AV Paclitaxel-Coated Percutaneous Transluminal Angioplasty (PTA) Balloon
- Standard Balloon Angioplasty: PTA was performed using a commercially available uncoated PTA balloon.
  Standard Balloon Angioplasty: Standard PTA Balloon
Arm/Group | IN.PACT AV DCB | Standard Balloon Angioplasty
Number analyzed (Participants) | 170 | 160
Percentage of participants
  3 Months | 91.4 | 84.6
  6 Months | 72.5 | 48.0
  9 Months | 66.8 | 43.1
  12 Months | 55.1 | 35.0
  18 Months | 43.6 | 28.8
  24 Months | 39.5 | 25.4
Statistical Analysis 1: Comparison: IN.PACT AV DCB vs Standard Balloon Angioplasty; Kaplan-Meier method was used to estimate access circuit primary patency; Test type: Superiority; p < 0.001, Log Rank — There is no planned hypothesis test other than at 6 months time point. P-value listed is at 6 months

4. Secondary Outcome: Target Lesion Primary Patency
Description: Percentage of participants with freedom from clinically driven target lesion revascularization or access thrombosis occurring in the target lesion through 3 months, 9 months,12 months, 18 months, and 24 months post-procedure.
Time Frame: 3, 9, 12, 18, and 24 Months
Population: There is no planned hypothesis test other than at 6 months time-point.
Measure: Number; unit: percentage of participants
Arm/Group | IN.PACT AV DCB | Standard Balloon Angioplasty
Number analyzed (Participants) | 170 | 160
percentage of participants
  3 Months | 96.9 | 90.3
  9 Months | 75.6 | 54.5
  12 Months | 65.3 | 46.3
  18 Months | 56.4 | 38.0
  24 Months | 52.2 | 36.2
Statistical Analysis 1: Comparison: IN.PACT AV DCB vs Standard Balloon Angioplasty; Kaplan-Meier method was used to estimate target lesion primary patency; Test type: Other — There is no planned hypothesis test other than at 6 months time point. P-value listed is at 6 months; p < 0.001, Log Rank — There is no planned hypothesis test other than at 6 months time point. P-value listed is at 6 months. Survival analysis was performed using Kaplan-Meier method; Survival analysis was performed using Kaplan-Meier method

5. Secondary Outcome: Cumulative Target Lesion Revascularizations
Description: The number and percentage of participants with target lesion revascularizations through 3 months, 6 months, 9 months,12 months, 18 months, and 24 months post-procedure.
Time Frame: 3, 6, 9,12, 18, and 24 Months
Population: Participants are included in the analyses up to the time consent was withdrawn, or they were exited, whichever is earlier.
Measure: Count of Participants; unit: Participants
Arm/Group | IN.PACT AV DCB | Standard Balloon Angioplasty
Number analyzed (Participants) | 170 | 160
Participants
  3 Months: number analyzed (Participants) | 160 | 155
  3 Months | 8 | 19
  6 Months: number analyzed (Participants) | 153 | 148
  6 Months | 25 | 59
  9 Months: number analyzed (Participants) | 147 | 144
  9 Months | 42 | 78
  12 Months: number analyzed (Participants) | 142 | 141
  12 Months | 57 | 88
  18 Months: number analyzed (Participants) | 134 | 136
  18 Months | 70 | 97
  24 Months: number analyzed (Participants) | 128 | 134
  24 Months | 76 | 101
Statistical Analysis 1: Comparison: IN.PACT AV DCB vs Standard Balloon Angioplasty; Test type: Superiority; p < 0.001, Chi-squared — There is no planned hypothesis test other than at 6 months time point. P-value listed is at 6 months

6. Secondary Outcome: Total Number of Interventions Required to Maintain Target Lesion Patency
Description: The number of target lesion revascularizations per treatment arm through 3 months, 6 months, 9 months, 12 months,18 months, and 24 months post-procedure.
Time Frame: 3, 6, 9, 12, 18, and 24 Months
Measure: Number; unit: Total number of interventions
Arm/Group | IN.PACT AV DCB | Standard Balloon Angioplasty
Number analyzed (Participants) | 170 | 160
Total number of interventions
  3 Months | 10 | 19
  6 Months | 32 | 70
  9 Months | 60 | 107
  12 Months | 93 | 144
  18 Months | 150 | 201
  24 Months | 193 | 235

7. Secondary Outcome: Total Number of Interventions Required to Maintain Access Circuit Patency
Description: The number of re-interventions in the target lesion and/or access circuit through 3 months, 6 months, 9 months,12 months, 18 months, and 24 months.
Time Frame: 3, 6, 9, 12, 18, and 24 Months
Measure: Number; unit: Total number of interventons
Arm/Group | IN.PACT AV DCB | Standard Balloon Angioplasty
Number analyzed (Participants) | 170 | 160
Total number of interventons
  3 Months | 16 | 23
  6 Months | 44 | 82
  9 Months | 74 | 124
  12 Months | 110 | 168
  18 Months | 180 | 248
  24 Months | 232 | 283

8. Secondary Outcome: Cumulative Access Circuit Thromboses
Description: The number and percentage of participants with access circuit thrombosis through 3 months, 6 months, 9 months, 12 months, 18 months, and 24 months.
Time Frame: 3, 6, 9, 12, 18, and 24 Months
Population: Participant withdrawn or lost-to-follow-up are included in the analyses up to the time consent was withdrawn, or they were exited, whichever is earlier.
Measure: Count of Participants; unit: Participants
Arm/Group | IN.PACT AV DCB | Standard Balloon Angioplasty
Number analyzed (Participants) | 170 | 160
Participants
  Access Circuit Thromboses Within 3 Months: number analyzed (Participants) | 160 | 155
  Access Circuit Thromboses Within 3 Months | 2 | 1
  Access Circuit Thromboses Within 6 Months: number analyzed (Participants) | 151 | 146
  Access Circuit Thromboses Within 6 Months | 3 | 5
  Access Circuit Thromboses Within 9 Months: number analyzed (Participants) | 146 | 143
  Access Circuit Thromboses Within 9 Months | 3 | 7
  Access Circuit Thromboses Within 12 Months: number analyzed (Participants) | 138 | 129
  Access Circuit Thromboses Within 12 Months | 4 | 8
  Access Circuit Thromboses Within 18 Months: number analyzed (Participants) | 126 | 119
  Access Circuit Thromboses Within 18 Months | 7 | 11
  Access Circuit Thromboses Within 24 Months: number analyzed (Participants) | 113 | 105
  Access Circuit Thromboses Within 24 Months | 7 | 13

9. Secondary Outcome: Device Success
Description: Device Success is defined as successful delivery, inflation, deflation and retrieval of the intact study balloon device without burst at or below rated burst pressure (RBP) during the index procedure.
Time Frame: Time of Procedure
Measure: Number; unit: Devices successfully used
Units Other Than Participants: Devices used
Arm/Group | IN.PACT AV DCB | Standard Balloon Angioplasty
Number analyzed (Participants) | 170 | 160
Number analyzed (Devices used) | 212 | 161
Devices successfully used | 212 | 161
Statistical Analysis 1: Comparison: IN.PACT AV DCB vs Standard Balloon Angioplasty; Test type: Superiority; p > 0.999, Chi-squared

10. Secondary Outcome: Procedure Success
Description: Maintenance of patency (≤30% residual stenosis) in the absence of peri-procedural serious adverse device effect (SADE).
Time Frame: Time of Procedure
Measure: Count of Participants; unit: Participants
Arm/Group | IN.PACT AV DCB | Standard Balloon Angioplasty
Number analyzed (Participants) | 170 | 160
Participants | 125 | 122
Statistical Analysis 1: Comparison: IN.PACT AV DCB vs Standard Balloon Angioplasty; Test type: Superiority; p = 0.482, Chi-squared

11. Secondary Outcome: Clinical Success
Description: Resumption of successful dialysis for at least one session after index procedure.
Time Frame: From the time of the index procedure to the first successful dialysis session after index procedure. Typically, this is within 1 week of index procedure.
Measure: Count of Participants; unit: Participants
Arm/Group | IN.PACT AV DCB | Standard Balloon Angioplasty
Number analyzed (Participants) | 159 | 154
Participants | 159 | 154
Statistical Analysis 1: Comparison: IN.PACT AV DCB vs Standard Balloon Angioplasty; Test type: Superiority; p > 0.999, Chi-squared

12. Secondary Outcome: Rate of Device Related Adverse Events
Description: Device Related Adverse Event Rate: defined as the number and percentage of participants with device related Adverse Events through 30 days, 3 months, 6 months, 9 months, 12 months, 18 months, and 24 months.
Time Frame: 30 days, 3, 6, 9, 12, 18, and 24 Months.
Population: Number of Participants with One or More Device-Related Adverse Events
Measure: Count of Participants; unit: Participants
Arm/Group | IN.PACT AV DCB | Standard Balloon Angioplasty
Number analyzed (Participants) | 170 | 160
Participants
  Subjects with device related AEs within 30 days | 2 | 2
  Subjects with device related AEs within 3 Months | 7 | 5
  Subjects with device related AEs within 6 Months | 10 | 7
  Subjects with device related AEs within 9 Months | 12 | 9
  Subjects with device related AEs within 12 Months | 12 | 9
  Subjects with device related AEs within 18 Months | 11 | 9
  Subjects with device related AEs within 24 Months | 11 | 9

13. Secondary Outcome: Procedure Related Adverse Event Rate
Description: Procedure Related Adverse Event Rate: defined as the number and percentage of participants with procedure related Adverse Events reported post-index procedure until the first successful dialysis session through 30 days, 3 months, 6 months, 9 months, 12 months, 18 months, and 24 months.
Time Frame: 30 Days, 3, 6, 9, 12, 18, and 24 Months
Population: Number of Participants with One or More Procedure-Related Adverse Events
Measure: Count of Participants; unit: Participants
Arm/Group | IN.PACT AV DCB | Standard Balloon Angioplasty
Number analyzed (Participants) | 170 | 160
Participants
  Subjects with Procedure-Related AEs within 30 Days | 7 | 7
  Subjects with Procedure-Related AEs within 3 Months | 7 | 7
  Subjects with Procedure-Related AEs within 6 Months | 7 | 7
  Subjects with Procedure-Related AEs within 9 Months | 8 | 8
  Subjects with Procedure-Related AEs within 12 Months | 8 | 8
  Subjects with Procedure-Related AEs within 18 Months | 8 | 8
  Subjects with Procedure-Related AEs within 24 Months | 8 | 8

14. Secondary Outcome: Target Lesion Revascularizations (TLR)
Description: Defined as the percentage of participants who had an event, the Kaplan-Meier method was used to estimate Cumulative Incidence up to 36 months post-index procedure.
Time Frame: 6, 9, 12, 18, 24, and 36 Months
Population: There is no planned hypothesis test.
Measure: Number; unit: % of Cumulative Incidence Rate
Arm/Group | IN.PACT AV DCB | Standard Balloon Angioplasty
Number analyzed (Participants) | 170 | 160
% of Cumulative Incidence Rate
  6 Months | 16.0 | 39.6
  9 Months | 27.8 | 53.1
  12 Months | 38.7 | 59.9
  18 Months | 48.4 | 66.3
  24 Months | 53.6 | 69.9
  36 Months | 62.5 | 79.3

15. Secondary Outcome: Clinically-Driven Target Lesion Revascularizations (CD-TLR)
Description: Defined as the percentage of participants who had an event, the Kaplan-Meier method was used to estimate Cumulative Incidence with CD-TLR up to 36 months post index procedure
Time Frame: 6, 9, 12, 18, 24, and 36 Months
Population: There is no planned hypothesis test for this endpoint.
Measure: Number; unit: Percentage of participants
Arm/Group | IN.PACT AV DCB | Standard Balloon Angioplasty
Number analyzed (Participants) | 170 | 160
Percentage of participants
  6 Months | 12.3 | 30.4
  9 Months | 23.4 | 44.8
  12 Months | 33.7 | 51.8
  18 Months | 42.7 | 60.1
  24 Months | 47.0 | 62.0
  36 Months | 54.9 | 69.1

16. Secondary Outcome: Re-interventions in the Access Circuit
Description: Defined as the percentage of participants who had a reinterventions occurring within the access circuit. The Kaplan-Meier method was used to estimate Cumulative Incidence up to 36 months post-index procedure.
Time Frame: 6, 9, 12, 18, 24, and 36 Months
Population: There is no planned hypothesis test for this endpoint.
Measure: Number; unit: Percentage of participants
Arm/Group | IN.PACT AV DCB | Standard Balloon Angioplasty
Number analyzed (Participants) | 170 | 160
Percentage of participants
  6 Months | 20.4 | 44.0
  9 Months | 32.2 | 56.8
  12 Months | 43.7 | 65.1
  18 Months | 55.6 | 70.8
  24 Months | 59.8 | 74.2
  36 Months | 71.9 | 83.1

17. Secondary Outcome: Abandonment of Target AVF
Description: Defined as number of participants with abandonment of the target AV up to 36 months post-index procedure.
Time Frame: 6, 9, 12, 18, 24, and 36 Months
Measure: Count of Participants; unit: Participants
Arm/Group | IN.PACT AV DCB | Standard Balloon Angioplasty
Number analyzed (Participants) | 170 | 160
Participants
  6 Months | 2 | 9
  9 Months | 3 | 10
  12 Months | 5 | 14
  18 Months | 13 | 18
  24 Months | 18 | 22
  36 Months | 23 | 25

18. Secondary Outcome: Serious Adverse Event Rate
Description: Serious Adverse Event Rate: defined as the number and percentage of participants with one or more Serious Adverse Events reported post-index procedure through 6 months, 12 months, 24 months, and 36 months.
Time Frame: 6, 12, 24, and 36 Months
Measure: Count of Participants; unit: Participants
Arm/Group | IN.PACT AV DCB | Standard Balloon Angioplasty
Number analyzed (Participants) | 170 | 160
Participants
  Subjects with SAEs within 180 Days | 71 | 85
  Subjects with SAEs within 360 Days | 105 | 115
  Subjects with SAEs within 720 Days | 131 | 128
  Subjects with SAEs within 1080 Days | 146 | 137

19. Secondary Outcome: Rate of Freedom From All-Cause Mortality Post Vital Status Update
Description: Percentage of participants who had all-cause death post vital status update. The Kaplan-Meier method was used to estimate survival probability up to 60 months post-index procedure through 6 months, 12 months, 24 months, 36 months, 48 months, and 60 months.
Time Frame: 6, 12, 24, 36, 48, and 60 Months
Measure: Number; unit: % of Survival
Arm/Group | IN.PACT AV DCB | Standard Balloon Angioplasty
Number analyzed (Participants) | 170 | 160
% of Survival
  Within 180 Days | 93.4 | 98.1
  Within 360 Days | 89.1 | 89.6
  Within 720 Days | 80.2 | 81.8
  Within 1080 Days | 73.4 | 68.8
  Within 1440 Days | 65.4 | 58.2
  Within 1800Days | 59.0 | 53.5

ADVERSE EVENTS:
Time Frame: All Adverse Events were collected from the time of consent through 6 Months post procedure. After 6 months, only SAEs, ADEs, SADEs, and UADEs were collected through 36 months. After 36 month, only vital status and SAEs related to death were collected and reported up to 60 months. Deaths in US participants who were alive at the time of discontinuing the study were collected and reported up to 60 months.
Description: All participant death within the database snapshot were included. Participants in the United States who were alive at the time of discontinuing the study continued to be monitored for death for up to 60 months. Any deaths that were observed in this population during this time period are included in the All-Cause Mortality data table. Events collected post vital update were included.
Arm/Group | IN.PACT AV DCB | Standard Balloon Angioplasty
All-Cause Mortality (participants affected / at risk) | 59/170 | 60/160
Serious Adverse Events (participants affected / at risk) | 148/170 | 143/160
Other Adverse Events (participants affected / at risk) | 31/170 | 32/160
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IN.PACT AV DCB (N=170) | Standard Balloon Angioplasty (N=160)
Anaemia (Blood and lymphatic system disorders) | 4 (5) | 3 (5)
Anaemia Of Chronic Disease (Blood and lymphatic system disorders) | 1 (2) | 0 (0)
Blood Loss Anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Coagulopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Nephrogenic Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Acute Coronary Syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Acute Left Ventricular Failure (Cardiac disorders) | 3 (5) | 0 (0)
Acute Myocardial Infarction (Cardiac disorders) | 3 (3) | 6 (6)
Angina Pectoris (Cardiac disorders) | 6 (9) | 6 (6)
Angina Unstable (Cardiac disorders) | 2 (2) | 0 (0)
Aortic Valve Incompetence (Cardiac disorders) | 1 (1) | 0 (0)
Aortic Valve Stenosis (Cardiac disorders) | 1 (1) | 2 (2)
Arteriosclerosis Coronary Artery (Cardiac disorders) | 0 (0) | 1 (1)
Atrial Fibrillation (Cardiac disorders) | 8 (8) | 5 (6)
Atrial Flutter (Cardiac disorders) | 4 (4) | 1 (1)
Atrioventricular Block (Cardiac disorders) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 2 (3) | 1 (1)
Cardiac Arrest (Cardiac disorders) | 8 (8) | 6 (7)
Cardiac Failure (Cardiac disorders) | 4 (4) | 1 (2)
Cardiac Failure Acute (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac Failure Chronic (Cardiac disorders) | 1 (2) | 2 (2)
Cardiac Failure Congestive (Cardiac disorders) | 8 (9) | 12 (14)
Cardio-Respiratory Arrest (Cardiac disorders) | 0 (0) | 1 (1)
Cardiogenic Shock (Cardiac disorders) | 0 (0) | 1 (1)
Cardiomyopathy (Cardiac disorders) | 2 (2) | 1 (2)
Chronic Left Ventricular Failure (Cardiac disorders) | 2 (2) | 0 (0)
Coronary Artery Disease (Cardiac disorders) | 6 (6) | 2 (2)
Coronary Artery Occlusion (Cardiac disorders) | 1 (1) | 0 (0)
Coronary Artery Stenosis (Cardiac disorders) | 4 (5) | 3 (3)
Diastolic Dysfunction (Cardiac disorders) | 1 (1) | 0 (0)
Ischaemic Cardiomyopathy (Cardiac disorders) | 2 (2) | 0 (0)
Mitral Valve Incompetence (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial Infarction (Cardiac disorders) | 0 (0) | 2 (2)
Myocardial Ischaemia (Cardiac disorders) | 2 (2) | 3 (3)
Pericardial Effusion (Cardiac disorders) | 3 (3) | 1 (1)
Pulseless Electrical Activity (Cardiac disorders) | 1 (1) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Acetylcholinesterase Deficiency (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Deafness Neurosensory (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Hyperparathyroidism Secondary (Endocrine disorders) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 4 (6) | 4 (4)
Glaucoma (Eye disorders) | 1 (1) | 0 (0)
Vitreous Haemorrhage (Eye disorders) | 1 (1) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
Ascites (Gastrointestinal disorders) | 2 (3) | 1 (1)
Colitis Ischaemic (Gastrointestinal disorders) | 1 (3) | 1 (2)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (2)
Diabetic Gastroparesis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 1 (1)
Diverticulum (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diverticulum Intestinal Haemorrhagic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 2 (2)
Faeces Discoloured (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric Polyps (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric Ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 3 (5) | 3 (5)
Gastrointestinal Necrosis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Inguinal Hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal Ischaemia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intra-Abdominal Haematoma (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ischaemic Enteritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Large Intestinal Stenosis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Large Intestine Polyp (Gastrointestinal disorders) | 1 (1) | 0 (0)
Lower Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Mesenteric Arterial Occlusion (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mesenteric Haematoma (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophageal Perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis Acute (Gastrointestinal disorders) | 0 (0) | 1 (1)
Portal Hypertensive Gastropathy (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectal Haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Small Intestinal Obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Upper Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 (1) | 2 (2)
Vomiting (Gastrointestinal disorders) | 2 (2) | 4 (4)
Asthenia (General disorders) | 1 (1) | 1 (1)
Chest Pain (General disorders) | 3 (3) | 5 (5)
Complication Associated With Device (General disorders) | 0 (0) | 1 (1)
Death (General disorders) | 18 (18) | 24 (24)
General Physical Health Deterioration (General disorders) | 1 (1) | 0 (0)
Multiple Organ Dysfunction Syndrome (General disorders) | 1 (1) | 0 (0)
Non-Cardiac Chest Pain (General disorders) | 0 (0) | 1 (1)
Peripheral Swelling (General disorders) | 0 (0) | 2 (2)
Physical Deconditioning (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 1 (1)
Stent-Graft Endoleak (General disorders) | 1 (1) | 0 (0)
Strangulated Hernia (General disorders) | 0 (0) | 1 (1)
Vascular Stent Occlusion (General disorders) | 1 (1) | 0 (0)
Vascular Stent Stenosis (General disorders) | 1 (2) | 2 (2)
Bile Duct Stone (Hepatobiliary disorders) | 1 (2) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 2 (2) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholecystitis Acute (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic Cirrhosis (Hepatobiliary disorders) | 1 (1) | 1 (1)
Hepatic Failure (Hepatobiliary disorders) | 1 (1) | 0 (0)
Kidney Transplant Rejection (Immune system disorders) | 0 (0) | 1 (1)
Abdominal Abscess (Infections and infestations) | 1 (1) | 0 (0)
Abscess Limb (Infections and infestations) | 2 (3) | 0 (0)
Acinetobacter Bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Anal Abscess (Infections and infestations) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Arteriovenous Fistula Site Infection (Infections and infestations) | 1 (2) | 0 (0)
Arteriovenous Graft Site Infection (Infections and infestations) | 0 (0) | 1 (1)
Arthritis Bacterial (Infections and infestations) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 2 (2) | 1 (1)
Bacterial Infection (Infections and infestations) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 3 (3) | 5 (5)
Cellulitis (Infections and infestations) | 7 (8) | 4 (4)
Clostridium Difficile Colitis (Infections and infestations) | 1 (1) | 1 (1)
Clostridium Difficile Infection (Infections and infestations) | 0 (0) | 1 (1)
Coronavirus Infection (Infections and infestations) | 2 (2) | 0 (0)
Covid-19 (Infections and infestations) | 4 (4) | 0 (0)
Covid-19 Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Cytomegalovirus Enteritis (Infections and infestations) | 1 (1) | 0 (0)
Device Related Infection (Infections and infestations) | 2 (4) | 0 (0)
Endocarditis (Infections and infestations) | 2 (2) | 0 (0)
Enterococcal Infection (Infections and infestations) | 0 (0) | 1 (1)
Escherichia Bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Escherichia Urinary Tract Infection (Infections and infestations) | 1 (1) | 0 (0)
Gangrene (Infections and infestations) | 5 (6) | 1 (1)
Gastroenteritis (Infections and infestations) | 4 (4) | 1 (1)
Gastrointestinal Infection (Infections and infestations) | 1 (1) | 0 (0)
Groin Infection (Infections and infestations) | 1 (1) | 0 (0)
Hordeolum (Infections and infestations) | 1 (1) | 0 (0)
Infected Dermal Cyst (Infections and infestations) | 1 (1) | 0 (0)
Infected Skin Ulcer (Infections and infestations) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 2 (2)
Influenza (Infections and infestations) | 6 (6) | 4 (5)
Intervertebral Discitis (Infections and infestations) | 1 (3) | 0 (0)
Klebsiella Bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Localised Infection (Infections and infestations) | 2 (2) | 0 (0)
Lower Respiratory Tract Infection (Infections and infestations) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Necrotising Fasciitis (Infections and infestations) | 0 (0) | 1 (1)
Osteomyelitis (Infections and infestations) | 6 (11) | 2 (4)
Peritonitis (Infections and infestations) | 0 (0) | 1 (2)
Pneumonia (Infections and infestations) | 19 (23) | 13 (15)
Pneumonia Aspiration (Infections and infestations) | 2 (2) | 2 (2)
Pneumonia Bacterial (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia Staphylococcal (Infections and infestations) | 0 (0) | 1 (1)
Portal Pyaemia (Infections and infestations) | 1 (1) | 0 (0)
Postoperative Wound Infection (Infections and infestations) | 0 (0) | 1 (1)
Pulmonary Sepsis (Infections and infestations) | 1 (1) | 1 (1)
Pustule (Infections and infestations) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 1 (1) | 1 (1)
Respiratory Syncytial Virus Infection (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 8 (8) | 6 (6)
Septic Shock (Infections and infestations) | 5 (5) | 1 (1)
Staphylococcal Bacteraemia (Infections and infestations) | 2 (3) | 2 (2)
Staphylococcal Infection (Infections and infestations) | 2 (4) | 0 (0)
Staphylococcal Osteomyelitis (Infections and infestations) | 1 (1) | 0 (0)
Staphylococcal Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Upper Respiratory Tract Infection (Infections and infestations) | 1 (1) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 3 (3) | 5 (6)
Urinary Tract Infection Bacterial (Infections and infestations) | 0 (0) | 1 (1)
Urosepsis (Infections and infestations) | 0 (0) | 1 (1)
Viral Infection (Infections and infestations) | 0 (0) | 2 (2)
Viral Upper Respiratory Tract Infection (Infections and infestations) | 1 (1) | 0 (0)
Wound Infection Staphylococcal (Infections and infestations) | 1 (1) | 0 (0)
Wound Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Acetabulum Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Anastomotic Stenosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ankle Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Arteriovenous Fistula Aneurysm (Injury, poisoning and procedural complications) | 9 (10) | 10 (11)
Arteriovenous Fistula Occlusion (Injury, poisoning and procedural complications) | 9 (19) | 20 (39)
Arteriovenous Fistula Site Complication (Injury, poisoning and procedural complications) | 86 (375) | 96 (427)
Arteriovenous Fistula Site Haematoma (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Arteriovenous Fistula Site Haemorrhage (Injury, poisoning and procedural complications) | 2 (2) | 3 (3)
Arteriovenous Fistula Site Pseudoaneurysm (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Arteriovenous Fistula Thrombosis (Injury, poisoning and procedural complications) | 6 (7) | 10 (12)
Arteriovenous Graft Site Pseudoaneurysm (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Arteriovenous Graft Site Stenosis (Injury, poisoning and procedural complications) | 1 (4) | 2 (6)
Burns Second Degree (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Complications Of Transplanted Kidney (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Coronary Artery Restenosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Femoral Neck Fracture (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Femur Fracture (Injury, poisoning and procedural complications) | 3 (3) | 1 (1)
Foot Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Haemodialysis Complication (Injury, poisoning and procedural complications) | 3 (3) | 1 (1)
Head Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hip Fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Humerus Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Inadequate Haemodialysis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Incarcerated Incisional Hernia (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Joint Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Limb Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Multiple Fractures (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Pelvic Fracture (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Radius Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Rectal Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Shunt Malfunction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Skull Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Spinal Compression Fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Subdural Haematoma (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Tibia Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Toxicity To Various Agents (Injury, poisoning and procedural complications) | 0 (0) | 2 (4)
Ulna Fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Upper Limb Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Vascular Access Malfunction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vascular Access Site Pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vascular Graft Complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vascular Graft Occlusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wound Dehiscence (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Anticoagulation Drug Level Below Therapeutic (Investigations) | 1 (1) | 0 (0)
Blood Pressure Decreased (Investigations) | 0 (0) | 1 (1)
Brain Natriuretic Peptide Increased (Investigations) | 1 (1) | 0 (0)
Occult Blood (Investigations) | 1 (1) | 0 (0)
Troponin Increased (Investigations) | 1 (1) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Failure To Thrive (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (2) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 7 (8) | 9 (11)
Hypernatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypervolaemia (Metabolism and nutrition disorders) | 6 (7) | 7 (8)
Hypoglycaemia (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
Hypovolaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Lactic Acidosis (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Malnutrition (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Type 2 Diabetes Mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Arthritis Reactive (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Chondrocalcinosis Pyrophosphate (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Costochondritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Flank Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Foot Deformity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Lumbar Spinal Stenosis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteolysis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Rheumatoid Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spinal Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spinal Stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Angiosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Bladder Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Breast Angiosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cholesteatoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Colon Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Hepatic Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastases To Peritoneum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Myelodysplastic Syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Parathyroid Tumour Benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Pituitary Tumour Benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Prostate Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Renal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Transitional Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0)
Amnesia (Nervous system disorders) | 0 (0) | 1 (1)
Aphasia (Nervous system disorders) | 0 (0) | 1 (1)
Brain Stem Stroke (Nervous system disorders) | 0 (0) | 1 (1)
Carotid Artery Stenosis (Nervous system disorders) | 0 (0) | 1 (1)
Carpal Tunnel Syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral Haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral Infarction (Nervous system disorders) | 1 (1) | 5 (5)
Cerebrovascular Accident (Nervous system disorders) | 4 (8) | 2 (2)
Cervical Radiculopathy (Nervous system disorders) | 0 (0) | 1 (1)
Cognitive Disorder (Nervous system disorders) | 1 (1) | 0 (0)
Cubital Tunnel Syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Dementia (Nervous system disorders) | 0 (0) | 1 (1)
Dementia Alzheimer's Type (Nervous system disorders) | 0 (0) | 1 (1)
Encephalopathy (Nervous system disorders) | 2 (2) | 3 (3)
Haemorrhagic Cerebral Infarction (Nervous system disorders) | 0 (0) | 1 (1)
Haemorrhagic Stroke (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Hepatic Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Hypertensive Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Ischaemic Stroke (Nervous system disorders) | 1 (1) | 1 (1)
Lacunar Infarction (Nervous system disorders) | 1 (1) | 0 (0)
Metabolic Encephalopathy (Nervous system disorders) | 2 (3) | 2 (3)
Myelopathy (Nervous system disorders) | 1 (1) | 0 (0)
Narcolepsy (Nervous system disorders) | 0 (0) | 1 (1)
Neuropathy Peripheral (Nervous system disorders) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 2 (3)
Spondylitic Myelopathy (Nervous system disorders) | 1 (1) | 1 (1)
Syncope (Nervous system disorders) | 2 (2) | 2 (4)
Thrombotic Cerebral Infarction (Nervous system disorders) | 0 (0) | 1 (1)
Toxic Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Transient Ischaemic Attack (Nervous system disorders) | 2 (5) | 0 (0)
Device Malfunction (Product Issues) | 1 (1) | 0 (0)
Confusional State (Psychiatric disorders) | 0 (0) | 1 (1)
Delirium Tremens (Psychiatric disorders) | 1 (1) | 0 (0)
Mental Status Changes (Psychiatric disorders) | 1 (1) | 6 (6)
Acute Kidney Injury (Renal and urinary disorders) | 1 (1) | 1 (1)
Chronic Kidney Disease (Renal and urinary disorders) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1)
End Stage Renal Disease (Renal and urinary disorders) | 2 (3) | 8 (8)
Haematuria (Renal and urinary disorders) | 1 (2) | 1 (1)
Renal Cyst (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal Failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal Mass (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary Retention (Renal and urinary disorders) | 0 (0) | 1 (1)
Benign Prostatic Hyperplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Acute Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 9 (15) | 6 (8)
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 5 (8) | 1 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 3 (5) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 6 (7) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary Hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (4)
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Respiratory Arrest (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 8 (10)
Acute Generalised Exanthematous Pustulosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Decubitus Ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dermal Cyst (Skin and subcutaneous tissue disorders) | 1 (3) | 0 (0)
Dermatitis Exfoliative Generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Diabetic Foot (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Erythema Multiforme (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Ischaemic Skin Ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin Mass (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin Ulcer (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Loss Of Personal Independence In Daily Activities (Social circumstances) | 1 (1) | 0 (0)
Refusal Of Treatment By Patient (Social circumstances) | 1 (1) | 0 (0)
Arteriovenous Fistula Operation (Surgical and medical procedures) | 2 (2) | 2 (2)
Cardiac Pacemaker Replacement (Surgical and medical procedures) | 1 (1) | 0 (0)
Dialysis Device Insertion (Surgical and medical procedures) | 0 (0) | 1 (1)
Intervertebral Disc Operation (Surgical and medical procedures) | 0 (0) | 1 (1)
Leg Amputation (Surgical and medical procedures) | 0 (0) | 1 (1)
Peripheral Revascularisation (Surgical and medical procedures) | 1 (1) | 0 (0)
Renal Transplant (Surgical and medical procedures) | 2 (2) | 1 (1)
Aneurysm (Vascular disorders) | 0 (0) | 1 (1)
Aortic Aneurysm (Vascular disorders) | 2 (2) | 0 (0)
Aortic Stenosis (Vascular disorders) | 2 (2) | 1 (1)
Arteriosclerosis (Vascular disorders) | 0 (0) | 1 (1)
Arteriovenous Fistula (Vascular disorders) | 1 (1) | 0 (0)
Brachiocephalic Vein Stenosis (Vascular disorders) | 1 (1) | 1 (1)
Deep Vein Thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Dry Gangrene (Vascular disorders) | 1 (1) | 0 (0)
Extremity Necrosis (Vascular disorders) | 1 (1) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 2 (2)
Haemorrhage (Vascular disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 2 (2) | 0 (0)
Hypertensive Crisis (Vascular disorders) | 1 (1) | 0 (0)
Hypertensive Emergency (Vascular disorders) | 2 (2) | 0 (0)
Hypertensive Urgency (Vascular disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 4 (4) | 6 (8)
Intermittent Claudication (Vascular disorders) | 1 (1) | 1 (1)
Peripheral Arterial Occlusive Disease (Vascular disorders) | 10 (15) | 8 (13)
Peripheral Artery Occlusion (Vascular disorders) | 1 (1) | 0 (0)
Peripheral Artery Stenosis (Vascular disorders) | 0 (0) | 2 (5)
Peripheral Ischaemia (Vascular disorders) | 2 (2) | 0 (0)
Peripheral Vascular Disorder (Vascular disorders) | 1 (1) | 0 (0)
Peripheral Vein Stenosis (Vascular disorders) | 2 (2) | 0 (0)
Secondary Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Shock Haemorrhagic (Vascular disorders) | 1 (1) | 0 (0)
Steal Syndrome (Vascular disorders) | 4 (5) | 4 (4)
Subclavian Artery Stenosis (Vascular disorders) | 1 (1) | 0 (0)
Subclavian Vein Occlusion (Vascular disorders) | 1 (3) | 0 (0)
Subclavian Vein Stenosis (Vascular disorders) | 1 (1) | 0 (0)
Subclavian Vein Thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Superior Vena Cava Stenosis (Vascular disorders) | 2 (2) | 0 (0)
Venous Stenosis (Vascular disorders) | 0 (0) | 2 (2)
Venous Thrombosis Limb (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IN.PACT AV DCB (N=170) | Standard Balloon Angioplasty (N=160)
Arteriovenous Fistula Site Complication (Injury, poisoning and procedural complications) | 31 (80) | 32 (128)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2022-01-20): https://cdn.clinicaltrials.gov/large-docs/67/NCT03041467/Prot_002.pdf
  • Statistical Analysis Plan (2022-02-07): https://cdn.clinicaltrials.gov/large-docs/67/NCT03041467/SAP_003.pdf